CLINICAL TRIAL: NCT05865964
Title: Evaluation of Anthropological, Socio-cultural and Psychological Factors of Surgeons Practising in Oncology Which Condition Brakes in the Evaluation of Surgical Innovations
Brief Title: Anthropological, Socio-cultural and Psychological Surgeons' Factors in Oncology and Brakes for Evaluation of Innovations
Acronym: SURGprofil
Status: Recruiting | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: West Cancerology Institute, France (Unknown); Toulouse Capitole University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22RD14
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Surgery
Keywords: Medical Care; clinical trial; innovation; breaks; surgeons; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The field of surgery continues to benefit from innovative solutions, changing surgical methods and techniques. Evaluation in terms of efficacy and Quality-Safety is an essential topic that directly affects the introduction of innovations. It is essential to carry out a robust evaluation strategy for surgical innovations, even if these are often opposed to drug innovations. The aim of this study is to investigate the anthropological, socio-cultural and psychological differences of surgeons that influence the evaluation of surgical innovations.

DETAILED DESCRIPTION:
RESEARCH HYPOTHESIS Over the past decade, the role of the surgeon in scientific research in oncology has evolved and many surgeons are involved in basic research activities alongside their clinical activities. Despite this increasing involvement in research, the issue of evaluation of surgical procedures remains a major concern. As an example, the French Society of Oncological Surgery programs at its annual congress a plenary session "Randomized trial: the grail in oncological surgery?". When the topic of clinical research is discussed, one of the first reactions is usually to point out the differences between research on new therapies and on surgical procedures. This persistent claim can be challenged. This claim may also be related to the major difference in regulation between therapeutics (MA) and medical devices (CE markings) which may not have encouraged surgeons to develop the culture of randomised evidence.

No study seems to evaluate the factors related to the surgeon influencing his involvement and participation in clinical research in oncological surgery. The aim of our study is to determine which anthropo-sociological factors in surgeons are associated with the obstacles to the evaluation of surgical innovations and influence their degree of participation in clinical research.

OBJECTIVES OF THE STUDY The main objective of this study is to evaluate the factors associated with the obstacles to the evaluation of surgical innovations.

The secondary objectives are :

* To identify the factors associated with involvement in clinical research on two levels : (i) Investigator coordinator, (ii) Investigator in a study.
* To assess knowledge of complementary designs to the randomised trial.
* To identify the parameters associated with 'knowledge' of the complementary regimens to the randomised trial.

STUDY DESIGN This is a prospective study conducted on a national scale in the form of a survey of surgeons working in cancerology. This project has obtained the support of UNICANCER (Federation of Cancer Centres), the French-speaking Society of Oncological Surgery (SFCO), the Head and Neck Tumour Study Group (GETTEC), the French Society of Cervico-facial Carcinology (SFCCF), French Society of Gynecology Oncology (SFOG), French Association of Digestive & Visceral Surgery and the French Society of Thoracic and Cardiovascular Surgery. Their mailings will be used to disseminate the survey to surgeons in the area.

STUDY PROCESS

Phase 1: Questionnaire creation

The first part of the project will consist in the creation of the questionnaire. The questionnaire will include data related to the surgeon (non-exhaustive list):

* Demography: age, gender
* Education :
* Place and date of graduation from medical school,
* Obtained DESC in oncology or European equivalent
* Practice :
* Speciality: senology, gynaecology,...
* Main place of practice: CHU, CLCC, CHG, Private clinic, ESPIC outside CLCC, Other,
* Number of treated patients per year.
* Involvement in clinical research:
* Accreditation to GCP Validated,
* Number of trials as Coordinating Investigator / Principal Investigator,
* Number of patients included in a clinical trial per year,
* Member of a learned society or cooperative group,

Questions associated with barriers to conducting trials in surgery and alternative methodological approaches will be drafted.

Practitioners' attitudes towards risk and uncertainty will be assessed by the following tools:

1. Questions on willingness to take risk in general and in different areas (answers given on a scale of 0-10).
2. Questions on the willingness to engage in risky activities in different areas (answers given on a scale of 0-10).
3. Choice of lotteries : choice between 6 lotteries characterised by different payoffs and risk levels.

In order to check the feasibility, the online questionnaire will be evaluated by the steering committee. The steering committee will include members from the sponsoring centre but also external members who will not be involved in the creation of the questionnaire. Once the questionnaire has been developed, the regulatory steps will be taken.

Phase 2: Awareness raising In this type of study, one of the key points is the response to the questionnaires. In order to mobilise a maximum of surgeons, actions (presentation, Webinar) will be carried out with the different groups/companies that have agreed to participate in the projects.

Phase 3: Sending of questionnaires The questionnaires will be sent to the different surgeons via the Sphynx survey software. This software allows the distribution of dynamic and interactive questionnaires with a display adapted to different media (computer, tablet, smartphone, etc.).

STATISTICAL METHODOLOGY Number of participants needed In two previous studies with a similar methodology, a response rate with usable questionnaires of 17 to 30% was observed, corresponding to 200 and 230 questionnaires. With 200 usable questionnaires and assuming that for 50% of them, obstacles to the evaluation of surgical innovations are identified, it is possible to carry out a multivariable model with 12 parameters according to the rule of thumb of 10 events per variable.

Statistical analysis Demographic data will be described by the usual descriptive statistics. Categorical variables will be presented as follows: number of missing data, number and percentage for each modality of the variable. Quantitative data will be presented as follows: median, minimum, maximum, number of missing data.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon practising oncology in France.
* E-mail address accessible via one of the companies/cooperating groups that have agreed to participate in the project

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgeon practising oncology in France.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Identification of the parameters associated with barriers to the evaluation of surgical innovations. | 21 months
  Logistic regression modelling will be carried out to identify the parameters associated with barriers to the evaluation of surgical innovations.
  The odds ratios will be estimated with their 95% confidence intervals. In accordance with the recommendations of the literature, a top-down stepwise procedure will be performed for the selection of variables.

SECONDARY OUTCOMES:
Identification of the parameters associated with involvement in clinical research. | 21 months
  Logistic regression modelling will be carried out to identify the parameters associated with involvement in clinical research.
  The odds ratios will be estimated with their 95% confidence intervals. In accordance with the recommendations of the literature, a top-down stepwise procedure will be performed for the selection of variables.
Identification of the parameters associated with knowledge of complementary patterns. | 21 months
  Knowledge of complementary patterns to the randomised trial will be presented using standard descriptive statistics. A similar strategy to the analysis of the primary objective will be used to identify parameters associated with knowledge of complementary patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bories P, Lamy S, Simand C, Bertoli S, Delpierre C, Malak S, Fornecker L, Moreau S, Recher C, Nebout A. Physician uncertainty aversion impacts medical decision making for older patients with acute myeloid leukemia: results of a national survey. Haematologica. 2018 Dec;103(12):2040-2048. doi: 10.3324/haematol.2018.192468. Epub 2018 Jul 13. PMID 30006448
- [Background] Brandberg Y, Malm M, Blomqvist L. A prospective and randomized study, "SVEA," comparing effects of three methods for delayed breast reconstruction on quality of life, patient-defined problem areas of life, and cosmetic result. Plast Reconstr Surg. 2000 Jan;105(1):66-74; discussion 75-6. doi: 10.1097/00006534-200001000-00011. PMID 10626972
- [Background] Castel P, Negrier S, Boissel JP; Plateforme d'Aide a la Recherche Clinique en Cancerologie de la region Rhone-Alpes. Why don't cancer patients enter clinical trials? A review. Eur J Cancer. 2006 Aug;42(12):1744-8. doi: 10.1016/j.ejca.2005.10.033. Epub 2006 Jun 14. PMID 16777404
- [Background] Concato J, Peduzzi P, Holford TR, Feinstein AR. Importance of events per independent variable in proportional hazards analysis. I. Background, goals, and general strategy. J Clin Epidemiol. 1995 Dec;48(12):1495-501. doi: 10.1016/0895-4356(95)00510-2. PMID 8543963
- [Background] Cook JA. The challenges faced in the design, conduct and analysis of surgical randomised controlled trials. Trials. 2009 Feb 6;10:9. doi: 10.1186/1745-6215-10-9. PMID 19200379
- [Background] Crocker JC, Farrar N, Cook JA, Treweek S, Woolfall K, Chant A, Bostock J, Locock L, Rees S, Olszowski S, Bulbulia R. Recruitment and retention of participants in UK surgical trials: survey of key issues reported by trial staff. BJS Open. 2020 Oct 4;4(6):1238-45. doi: 10.1002/bjs5.50345. Online ahead of print. PMID 33016008
- [Background] Cros F, Lamy S, Grosclaude P, Nebout A, Chabrillac E, Vergez S, Bories P, Dupret-Bories A. Physician practice variation in head and neck cancer therapy: Results of a national survey. Oral Oncol. 2021 Jun;117:105293. doi: 10.1016/j.oraloncology.2021.105293. Epub 2021 Apr 14. PMID 33862559
- [Background] Elliott D, Hamdy FC, Leslie TA, Rosario D, Dudderidge T, Hindley R, Emberton M, Brewster S, Sooriakumaran P, Catto JWF, Emara A, Ahmed H, Whybrow P, le Conte S, Donovan JL. Overcoming difficulties with equipoise to enable recruitment to a randomised controlled trial of partial ablation vs radical prostatectomy for unilateral localised prostate cancer. BJU Int. 2018 Dec;122(6):970-977. doi: 10.1111/bju.14432. Epub 2018 Aug 15. PMID 29888845
- [Background] Evrard S, McKelvie-Sebileau P, van de Velde C, Nordlinger B, Poston G. What can we learn from oncology surgical trials? Nat Rev Clin Oncol. 2016 Jan;13(1):55-62. doi: 10.1038/nrclinonc.2015.176. Epub 2015 Oct 20. PMID 26483296
- [Background] Filleron T, Bonnetain F, Mancini J, Martinez A, Roche H, Dalenc F. Prospective construction and validation of a prognostic score to identify patients who benefit from third-line chemotherapy for metastatic breast cancer in terms of overall survival: the METAL3 Study. Contemp Clin Trials. 2015 Jan;40:1-8. doi: 10.1016/j.cct.2014.11.005. Epub 2014 Nov 8. PMID 25460338
- [Background] Filleron T, Lusque A, Dalenc F, Ferron G, Roche H, Martinez A, Jouve E. Alternative methodological approach to randomized trial for surgical procedures routinely used. Contemp Clin Trials. 2018 May;68:109-115. doi: 10.1016/j.cct.2018.03.016. Epub 2018 Mar 30. PMID 29608972
- [Background] Fisher B, Montague E, Redmond C, Barton B, Borland D, Fisher ER, Deutsch M, Schwarz G, Margolese R, Donegan W, Volk H, Konvolinka C, Gardner B, Cohn I Jr, Lesnick G, Cruz AB, Lawrence W, Nealon T, Butcher H, Lawton R. Comparison of radical mastectomy with alternative treatments for primary breast cancer. A first report of results from a prospective randomized clinical trial. Cancer. 1977 Jun;39(6 Suppl):2827-39. doi: 10.1002/1097-0142(197706)39:63.0.co;2-i. No abstract available. PMID 326381
- [Background] Ford E, Jenkins V, Fallowfield L, Stuart N, Farewell D, Farewell V. Clinicians' attitudes towards clinical trials of cancer therapy. Br J Cancer. 2011 May 10;104(10):1535-43. doi: 10.1038/bjc.2011.119. Epub 2011 Apr 12. PMID 21487408
- [Background] Giuliano AE, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Hunt KK, Morrow M, Ballman K. Locoregional recurrence after sentinel lymph node dissection with or without axillary dissection in patients with sentinel lymph node metastases: the American College of Surgeons Oncology Group Z0011 randomized trial. Ann Surg. 2010 Sep;252(3):426-32; discussion 432-3. doi: 10.1097/SLA.0b013e3181f08f32. PMID 20739842
- [Background] Goyal A, Dodwell D. POSNOC: A Randomised Trial Looking at Axillary Treatment in Women with One or Two Sentinel Nodes with Macrometastases. Clin Oncol (R Coll Radiol). 2015 Dec;27(12):692-5. doi: 10.1016/j.clon.2015.07.005. Epub 2015 Aug 5. No abstract available. PMID 26254841
- [Background] Goyal A, Mann GB, Fallowfield L, Duley L, Reed M, Dodwell D, Coleman RE, Fakis A, Newcombe R, Jenkins V, Whitham D, Childs M, Whynes D, Keeley V, Ellis I, Fairbrother P, Sadiq S, Monson K, Montgomery A, Tan W, Vale L, Homer T, Badger H, Haines RH, Lewis M, Megias D, Nabi Z, Singh P, Caraman A, Miles E; POSNOC Trialists. POSNOC-POsitive Sentinel NOde: adjuvant therapy alone versus adjuvant therapy plus Clearance or axillary radiotherapy: a randomised controlled trial of axillary treatment in women with early-stage breast cancer who have metastases in one or two sentinel nodes. BMJ Open. 2021 Dec 2;11(12):e054365. doi: 10.1136/bmjopen-2021-054365. PMID 34857578
- [Background] Gray S, Price C. Barriers to participation in randomised controlled trials. J Clin Epidemiol. 2001 Mar;54(3):323-4. doi: 10.1016/s0895-4356(00)00279-1. No abstract available. PMID 11243239
- [Background] Halsted WS. I. A Clinical and Histological Study of certain Adenocarcinomata of the Breast: and a Brief Consideration of the Supraclavicular Operation and of the Results of Operations for Cancer of the Breast from 1889 to 1898 at the Johns Hopkins Hospital. Ann Surg. 1898 Nov;28(5):557-76. No abstract available. PMID 17860646
- [Background] Hirst A, Agha RA, Rosin D, McCulloch P. How can we improve surgical research and innovation?: the IDEAL framework for action. Int J Surg. 2013;11(10):1038-42. doi: 10.1016/j.ijsu.2013.09.016. Epub 2013 Oct 7. No abstract available. PMID 24113195
- [Background] Jones RP, Are C, Hugh TJ, Grunhagen DJ, Xu J, Balch CM, Poston GJ. Reshaping the critical role of surgeons in oncology research. Nat Rev Clin Oncol. 2019 May;16(5):327-332. doi: 10.1038/s41571-018-0149-1. PMID 30617343
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876
- [Background] McLeod RS. Issues in surgical randomized controlled trials. World J Surg. 1999 Dec;23(12):1210-4. doi: 10.1007/s002689900649. PMID 10552108
- [Background] Mishra-Kalyani PS, Amiri Kordestani L, Rivera DR, Singh H, Ibrahim A, DeClaro RA, Shen Y, Tang S, Sridhara R, Kluetz PG, Concato J, Pazdur R, Beaver JA. External control arms in oncology: current use and future directions. Ann Oncol. 2022 Apr;33(4):376-383. doi: 10.1016/j.annonc.2021.12.015. Epub 2022 Jan 10. PMID 35026413
- [Background] Moons KG, Altman DG, Reitsma JB, Ioannidis JP, Macaskill P, Steyerberg EW, Vickers AJ, Ransohoff DF, Collins GS. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): explanation and elaboration. Ann Intern Med. 2015 Jan 6;162(1):W1-73. doi: 10.7326/M14-0698. PMID 25560730
- [Background] Nakamura S. Axillary lymph node dissection in sentinel node positive breast cancer: is it necessary? Curr Opin Obstet Gynecol. 2013 Feb 19. doi: 10.1097/GCO.0b013e32834f3608. Online ahead of print. PMID 23425664
- [Background] Potter S, Mills N, Cawthorn SJ, Donovan J, Blazeby JM. Time to be BRAVE: is educating surgeons the key to unlocking the potential of randomised clinical trials in surgery? A qualitative study. Trials. 2014 Mar 14;15:80. doi: 10.1186/1745-6215-15-80. PMID 24628821
- [Background] Ross S, Grant A, Counsell C, Gillespie W, Russell I, Prescott R. Barriers to participation in randomised controlled trials: a systematic review. J Clin Epidemiol. 1999 Dec;52(12):1143-56. doi: 10.1016/s0895-4356(99)00141-9. PMID 10580777
- [Background] Schroen AT, Brenin DR. Breast cancer treatment beliefs and influences among surgeons in areas of scientific uncertainty. Am J Surg. 2010 Apr;199(4):491-9. doi: 10.1016/j.amjsurg.2009.04.005. PMID 20359569
- [Background] Spillane AJ, Mann GB. Surgeon knows best versus breast cancer surgical clinical trial equipoise: a plea for the sake of future trials. ANZ J Surg. 2017 Mar;87(3):111-112. doi: 10.1111/ans.13831. No abstract available. PMID 28253558
- [Background] Taylor KM, Margolese RG, Soskolne CL. Physicians' reasons for not entering eligible patients in a randomized clinical trial of surgery for breast cancer. N Engl J Med. 1984 May 24;310(21):1363-7. doi: 10.1056/NEJM198405243102106. PMID 6717508
- [Background] Tibau A, Molto C, Borrell M, Del Paggio JC, Barnadas A, Booth CM, Amir E. Magnitude of Clinical Benefit of Cancer Drugs Approved by the US Food and Drug Administration Based on Single-Arm Trials. JAMA Oncol. 2018 Nov 1;4(11):1610-1611. doi: 10.1001/jamaoncol.2018.4300. PMID 30267037
- [Background] Tolaney SM, Barry WT, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis M, Shapira I, Wolff AC, Carey LA, Overmoyer BA, Partridge AH, Guo H, Hudis CA, Krop IE, Burstein HJ, Winer EP. Adjuvant paclitaxel and trastuzumab for node-negative, HER2-positive breast cancer. N Engl J Med. 2015 Jan 8;372(2):134-41. doi: 10.1056/NEJMoa1406281. PMID 25564897
- [Background] Unger JM, Hershman DL, Till C, Minasian LM, Osarogiagbon RU, Fleury ME, Vaidya R. "When Offered to Participate": A Systematic Review and Meta-Analysis of Patient Agreement to Participate in Cancer Clinical Trials. J Natl Cancer Inst. 2021 Mar 1;113(3):244-257. doi: 10.1093/jnci/djaa155. PMID 33022716